CLINICAL TRIAL: NCT01926587
Title: A Phase I/II, Multi-center, Dose-escalating Study of the Tolerability, Pharmacokinetics, and Clinical Activity of the Combined Administration of Oral Rigosertib With Azacitidine in Patients With Myelodysplastic Syndrome or Acute Myeloid Leukemia
Brief Title: Phase II Part 2 Expansion of Oral Rigosertib in Combination With Azacitidine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Onconova 09-08; 2013-000673-72 (EudraCT Number)
Record Dates: First submitted 2013-08-18; First posted 2013-08-21 (Estimated); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Myelodysplastic Syndrome; Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia
Keywords: rigosertib; ON 01910.Na; azacitidine; Vidaza
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic | interventions — ON 01910; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral rigosertib plus azacitidine (Experimental): Oral rigosertib will be administered twice a day in fasting conditions for weeks 1, 2, and 3 of a 4-week cycle. Starting on Day 1 of second week (Day 8) of the cycle, azacitidine will be administered by subcutaneous injection or intravenous infusion at the labeled daily dose of 75 mg/m2, for 7 days.
  Interventions: Drug: oral rigosertib; Drug: Azacitidine

INTERVENTIONS:
Drug: oral rigosertib — Oral rigosertib will be administered twice a day in fasting conditions for weeks 1, 2, and 3 of a 4-week cycle.
  Other Names: ON 01910.Na
Drug: Azacitidine — Starting on Day 1 of second week (Day 8) of the cycle, azacitidine will be administered by subcutaneous injection or intravenous infusion at the labeled daily dose of 75 mg/m2, for 7 days.
  Other Names: Vidaza

SUMMARY:
This study, is a Phase I/II clinical trial in three parts: Phase I Dose Escalation, Phase II, Part 1 RPTD Cohort, and Phase II, Part 2 Expansion. The first two parts have been completed. The Phase II, Part 2 Expansion will assess if treatment with rigosertib in combination with azacitidine, has measurable effects in patients with myelodysplastic syndrome (MDS). Safety of patients is an objective throughout all parts of the study.

DETAILED DESCRIPTION:
This will be a Phase I/II open-label, single-arm, dose-escalating, multicenter study, in three parts: Phase I Dose Escalation, Phase II, Part 1 RPTD Cohort, and Phase II, Part 2 Expansion, in which patients with myelodysplastic syndrome (MDS), acute myeloid leukemia (AML), or chronic myelomonocytic leukemia (CMML) will receive subcutaneous (SC) or intravenous (IV) azacitidine per approved label in combination with oral rigosertib. The first two parts of the study have been completed.

The Phase II Part 2 Expansion will enroll up to 40 patients, randomized 1:1 into 2 cohorts of up to 20 patients each, to receive 1120 mg of rigosertib over 24 hours: either 560 mg in the morning and 560 mg in the afternoon, or 840 mg in the morning and 280 mg in the afternoon. The afternoon dose in both cohorts must be administered at 3 PM (±1 hr) at least 2 hr after lunch. In the Phase II, Part 2 Expansion patients with RAEB t/non-proliferative AML will be eligible, however patients with CMML will not.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MDS, CMML, or RAEB-t/non-proliferative AML (as defined by 20-30% BMBL, WBC ≤ 25,000 x 10^9/L and stable for at least 4 weeks without intervention) according to World Health Organization (WHO) criteria or French American British (FAB) classification either previously treated or previously untreated. The diagnosis must be confirmed via BM aspirate and/or biopsy within 6 weeks prior to Screening. Note: patients with RAEB-t/non-proliferative AML (as defined by 20-30% BMBL, WBC ≤ 25,000 x 10^9/L and stable for at least 4 weeks without intervention) are not eligible for the Phase II Part 1 RPTD component of the study and patients with CMML will not be eligible for Phase II Part 2 Expansion of the study.
* If the patient has been diagnosed with MDS, disease of patient must be classified as Int-1, Intermediate-2 (Int-2) or High-risk, according to International Prognosis Scoring System (IPSS) classification. Note: Only Int-2 or High-risk patients will be enrolled at French site.
* Off all other treatments for MDS, CMML, or AML including an erythropoiesis-stimulating agent (ESA), for at least 4 weeks prior to Screening. Filgrastim (G-CSF) is allowed before and during the study, as clinically indicated.
* For AML patients, no more than 1 prior salvage therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
* Willing to adhere to the prohibitions and restrictions specified in this protocol.
* The patient must signed an informed consent form indicating that she/he understands the purpose of and procedures required for the study and is willing to participate in the study.

Exclusion Criteria:

* Prior treatment with rigosertib;
* Anemia due to factors other than MDS, CMML, or AML (including hemolysis or gastrointestinal bleeding).
* Any active malignancy within the past year, except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix or breast.
* Uncontrolled intercurrent illness.
* Active infection not adequately responding to appropriate therapy.
* Total bilirubin ≥ 2.0 mg/dL not related to Gilbert's disease or hemolysis.
* Alanine transaminase (ALT)/aspartate transaminase (AST) ≥ 2.5 x upper limit of normal (ULN).
* Serum creatinine ≥ 2.0 mg/dL.
* Ascites requiring active medical management including paracentesis.
* Hyponatremia (defined as serum sodium value of < 130 mEq/L).
* Female patients who are pregnant or lactating.
* Female patients of childbearing potential and male patients with partners of childbearing potential who are unwilling to follow strict contraception requirements before entry and throughout the study, up to and including the 30-day nontreatment follow-up period.
* Female patients with reproductive potential who do not have a negative blood or urine pregnancy test at Screening.
* Major surgery without full recovery or major surgery within 3 weeks of Screening.
* Uncontrolled hypertension (defined as a systolic pressure ≥ 160 mmHg and/or a diastolic pressure ≥ 110 mmHg).
* New onset seizures (within 3 months prior to Screening) or poorly controlled seizures.
* Any other investigational agent or chemotherapy, radiotherapy, or immunotherapy administered within 4 weeks prior to Screening.
* Chronic use (˃ 2 weeks) of corticosteroids (˃ 10 mg/24 hr equivalent prednisone) within 4 weeks of Baseline/First Dose.
* Investigational therapy within 4 weeks of Screening.
* Psychiatric illness or social situation that would limit the patient's ability to tolerate and/or comply with study requirements.
* Patients with RAEB-t/non-proliferative AML (as defined by 20-30% BMBL, WBC ≤ 25,000 x 10^9/L and stable for at least 4 weeks without intervention) are not eligible to participate in the Phase II Part 1 RPTD component of the study and patients with CMML will not be eligible for Phase II Part 2 of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-08; Primary Completion 2020-12-08 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
Dose escalation part of study: Number of patients in whom Dose a Limiting Toxicity (DLT) are observed | 28 days
  Dose Limiting Toxicity is defined as Grade 3 or greater non-hematological toxicity or stomatitis and/or esophagitis/dysphagitis lasting longer than 3 days.
Dose escalation part of study: Number of patients in whom adverse events are observed | Up to 48 weeks
  Adverse events will be coded using the most recent version of the Medical Dictionary for Regulatory Activities (MedDRA) and summarized by system organ class (SOC), preferred term (PT), and worst Common Terminology Criteria for Adverse Events (CTCAE) Version 4 grade per patient.
In Phase 2 of study: Number of patients in whom adverse events are observed | Up to 48 weeks
  Adverse events will be coded using the most recent version of the Medical Dictionary for Regulatory Activities (MedDRA) and summarized by system organ class (SOC), preferred term (PT), and worst Common Terminology Criteria for Adverse Events (CTCAE) Version 4 grade per patient.
In Phase 2 of study: Area Under the Curve (AUC) | Day 1 and Day 15
  The following time points will be used to collect samples to determine the AUC on Day 1 and 15: Pre-dose the first dose of the day and at 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, and 8.0 hour post dose the first dose of the day.
In Phase 2 of the study: Cmax | Days 1 and 15.
  The following time points will be used to collect samples to determine the Cmax on Day 1 and 15: Pre-dose the first dose of the day and at 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, and 8.0 hour post dose the first dose of the day.

SECONDARY OUTCOMES:
Number of patients with complete or partial response | Up to 48 weeks
  Complete remission (CR) or partial remission (PR) or bone marrow CR according to 2006 International Working Group criteria.
Number of patients in whom improvements in absolute neutrophil count, platelet count, and erythroid responses are observed | Up to 48 weeks.
  Hematologic Improvement according to 2006 International Working Group criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Steven M. Fruchtman, MD, Study Chair — Traws Pharma, Inc.
Locations (13):
- United States (12):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope, Duarte, California
  - Desert Hematology Oncology Medical Group, Inc., Rancho Mirage, California
  - Rush University Medical Center, Chicago, Illinois
  - Cancer Center of Kansas, Wichita, Kansas
  - Saint Louis University, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai Medical Center, New York, New York
  - White Plains Hospital Center for Cancer Care, White Plains, New York
  - Carolina Blood and Cancer Care Associates, Rock Hill, South Carolina
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Hôpital St. Louis, Paris, France

REFERENCES:
- [Background] Navada SC, Silverman LR. The safety and efficacy of rigosertib in the treatment of myelodysplastic syndromes. Expert Rev Anticancer Ther. 2016 Aug;16(8):805-10. doi: 10.1080/14737140.2016.1209413. Epub 2016 Jul 15. PMID 27400247
- [Background] Chaurasia, P. et al. Rigosertib in Combination with Azacitidine Modulates Epigenetic Pathways and can Overcome Clinical Resistance to Hypomethylating Agents in Myelodysplastic Syndromes (MDS). Leukemia Research , Volume 55 , S121, April 2017; MDS 2017.
- [Result] Garcia-Manero G, Fenaux P. Comprehensive Analysis of Safety: Rigosertib in 557 Patients with Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML). Blood Dec 2016, 128 (22) 2011; ASH 2016.
- [Result] Navada S, Garcia-Manero G. Combination of Oral Rigosertib and Injectable Azacitidine in Patients with Myelodysplastic Syndromes (MDS): Results from a Phase II Study. Blood Dec 2016, 128 (22) 3167; ASH 2016.
- [Result] Navada, S. et al. Combination of Oral Rigosertib and Injectable Azacitidine in Patients with Myelodysplastic Syndromes (MDS). Leukemia Research , Volume 55 , S30, April 2017; MDS 2017.
- [Derived] Navada SC, Garcia-Manero G, OdchimarReissig R, Pemmaraju N, Alvarado Y, Ohanian MN, John RB, Demakos EP, Zbyszewski PS, Maniar M, Woodman RC, Fruchtman SM, Silverman LR. Rigosertib in combination with azacitidine in patients with myelodysplastic syndromes or acute myeloid leukemia: Results of a phase 1 study. Leuk Res. 2020 Jul;94:106369. doi: 10.1016/j.leukres.2020.106369. Epub 2020 May 12. PMID 32442785
- See also: Information about clinical trials at MD Anderson Cancer Center — http://www.mdanderson.org/patient-and-cancer-information/cancer-information/clinical-trials/clinical-trials-at-md-anderson/index.html